CLINICAL TRIAL: NCT06088043
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo- and Active Comparator-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-279 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study About How Well TAK-279 Works and Its Safety in Participants With Moderate-to-severe Plaque Psoriasis During 52 Weeks of Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-3001; jRCT2031230583 (Registry Identifier: jRCT); 2023-505841-22-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis
Keywords: Drug Therapy; Latitude Psoriasis 1, Latitude Research Program
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-279 (Experimental)
  Interventions: Drug: TAK-279
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Apremilast (Active Comparator)
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: TAK-279 — Specified drug on specified days.
  Arms: TAK-279
Drug: Placebo — Specified drug on specified days.
  Arms: Placebo
Drug: Apremilast — Specified drug on specified days.
  Arms: Apremilast

SUMMARY:
The main aim of this study is to show how well TAK-279 reduces the skin plaques compared to placebo, in participants with moderate-to-severe plaque psoriasis. Participants will be assigned to one of the 3 study treatments (TAK-279, apremilast (an approved treatment), or a placebo). Participants will be in the study for up to 61 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. TAK-279 is being tested to treat people with moderate to severe plaque psoriasis.

The study will enroll approximately 600 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the following treatment groups in a ratio of 3:1:1 to receive TAK-279, placebo, or apremilast which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

1. TAK-279
2. Placebo
3. Apremilast

This multi-center trial will be conducted worldwide. Participants will go through a screening process to make sure they meet the rules for taking part in the study. This will take up to 35 days. If participants meet the study rules, they will be treated for up to 52 weeks (1 year). There will be a safety follow-up visit 4 weeks after their last day of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Plaque psoriasis for at least 6 months.
2. Moderate to severe disease.
3. Candidate for phototherapy or systemic therapy.

Exclusion Criteria:

1. Other forms of psoriasis.
2. History of recent infection.
3. Prior exposure to TAK-279 or active comparator.

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving >=75% Improvement from Baseline in Psoriasis Area and Severity Index (PASI) Score (PASI-75 Response) at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving 90% Improvement from Baseline in PASI (PASI-90 Response) at Week 16 Comparing TAK-279 Against Placebo | Baseline, Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. Higher scores indicate worsening. 'Clear' will include all participants who score a 0.
Percentage of Participants Achieving PASI-100 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving a Scalp-specific Physician's Global Assessment (ssPGA) of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants with a Baseline Dermatology Life Quality Index (DLQI) Score >=2 who Achieve DLQI Score of 0 or 1 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's quality of life (QoL) during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants with a Baseline Psoriasis Symptoms and Signs Diary (PSSD) >=1 who Achieve Weekly Mean PSSD Symptom Score of 0 at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in Nail Psoriasis Severity Index (NAPSI) at Week 16 Among Participants with Nail Involvement at Baseline Comparing TAK-279 Against Placebo | Baseline and Week 16
  The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each nail will be scored for both nail matrix and nail bed psoriasis for each quadrant (ranging from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores indicate more severe psoriasis.
Change from Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percent Change from Baseline in Body Surface Area (BSA) Affected by Psoriasis at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage of Participants Achieving a Physician's Global Assessment (PGA) of the Hands and/or Feet of Clear (0) or Almost Clear (1) with a >=2-Point Decrease From Baseline at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  PGA is a 5-point scale and a score of 0 to 4 should be assigned, based on the category that best describes the severity of active psoriasis of the participant's hands and/or feet (palmoplantar), where 0=clear and 4=severe. Higher scores indicate worsening of severity. It will be evaluated for participants with the presence of active hand or foot psoriasis on Day 1.
Change from Baseline in DLQI at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life). It will be evaluated for participants with a baseline DLQI score >=2.
Change from Baseline in the Short Form-36 Health Survey (SF-36) Version 2 Scores at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  The SF-36 is a self-administered, validated questionnaire designed to measure generic health-related QoL. This 36-item questionnaire measures 8 domains, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Two summary scores, including the physical component summary (PCS) and mental component summary (MCS), will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL.
Change from Baseline in the EuroQoL 5-Dimension 5-level Questionnaire (EQ-5D-5L) Scores at Week 16 Comparing TAK-279 Against Placebo | Baseline and Week 16
  EQ-5D-5L includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 response levels for each domain (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). The scores in the 5 dimensions will be summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health; 0=a health state equivalent to death, and 1=perfect health.
Change in Work Productivity and Activity Impairment-Psoriasis (WPAI-PSO) Questionnaire Scores at Week 16 Comparing TAK-279 Against Placebo | Week 16
  The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and impairment in activities performed outside of work. Each WPAI score will be expressed as impairment percentages (0-100) with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Apremilast | Baseline and Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. Higher scores indicate worsening. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 24 Comparing TAK-279 Against Apremilast | Baseline and Week 24
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Change from Baseline in Weekly Mean PSSD Symptom Score at Week 16 Comparing TAK-279 Against Apremilast | Baseline and Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Percentage of Participants Achieving an ssPGA of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving PASI-100 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-100 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing 100% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants with a Baseline DLQI Score >=2 who Achieve DLQI Score of 0/1 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants with a Baseline PSSD >=1 who Achieve a Weekly Mean PSSD Symptom Score of 0 at Week 16 Comparing TAK-279 Against Apremilast | Week 16
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in NAPSI, Among Participants with Nail Involvement at Baseline at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each nail will be scored for both nail matrix and nail bed psoriasis for each quadrant (ranging from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores indicate more severe psoriasis.
Percentage of Participants Achieving an ssPGA of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Week 24 Comparing TAK-279 Against Apremilast | Baseline and Week 24
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Change from Baseline in DLQI at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Change from Baseline in BSA Affected by Psoriasis at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percent Change from Baseline in BSA Affected by Psoriasis at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  Psoriasis BSA will be assessed by means of the handprint method, where the surface of the palm and 5 digits of the participant's hand represents 1% BSA. The sum of handprints equates to the total surface area of involvement.
Percentage of Participants Achieving an sPGA of Clear (0) at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' will include all participants who score a 0.
Percentage of Participants with a Baseline DLQI Score >=2 who Achieve a DLQI Score of 0/1 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicate: 0-1 (no effect on participant's life), 2-5 (small effect on participant's life), 6-10 (moderate effect on participant's life), 11-20 (very large effect on participant's life), 21-30 (extremely large effect on participant's life).
Percentage of Participants with a Baseline PSSD >=1 who Achieve a Weekly Mean PSSD Symptom Score of 0 at Week 24 Comparing TAK-279 Against Apremilast | Week 24
  The PSSD is an 11-item validated questionnaire that assesses symptoms (itch, pain, stinging, burning, and skin tightness) and participant-observable signs (skin dryness, cracking, scaling, shedding/flaking, redness, and bleeding) of moderate-to-severe plaque psoriasis. These symptoms and signs will be evaluated by asking participants to assign a numerical score representing of worst intensity over the last 24-hour on a scale from 0 to 10, with 0 indicating absence of symptoms or signs and 10 indicating worst imaginable symptoms or signs. The PSSD is a composite score calculated based on the scores for each question that can range between 0 and 100. A higher score indicates more severe disease.
Change from Baseline in ssPGA at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  ssPGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Percentage of Participants Achieving a PGA of the Hands and/or Feet of Clear (0) or Almost Clear (1) with a >=2-Point Decrease From Baseline at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  PGA is a 5-point scale and a score of 0 to 4 should be assigned, based on the category that best describes the severity of active psoriasis of the participant's hands and/or feet (palmoplantar), where 0=clear and 4=severe. Higher scores indicate worsening of severity. It will be evaluated for participants with the presence of active hand or foot psoriasis on Day 1.
Change from Baseline in SF-36 Version 2 Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The SF-36 is a self-administered, validated questionnaire designed to measure generic health-related QoL. This 36-item questionnaire measures 8 domains, including physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health, physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Two summary scores, including the PCS and MCS, will be calculated ranging from 0 (worst) to 100 (best). Higher scores indicate better QoL.
Change from Baseline in the EQ-5D-5L Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  EQ-5D-5L includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 response levels for each domain (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). The scores in the 5 dimensions will be summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health; 0=a health state equivalent to death, and 1=perfect health.
Change from Baseline in the WPAI-PSO Scores at Weeks 16 and 24 Comparing TAK-279 Against Apremilast | Baseline, Weeks 16 and 24
  The WPAI-PSO consists of 6 questions to determine employment status, hours missed from work because of psoriasis, hours missed from work for other reasons, hours actually worked, the degree to which psoriasis affected work productivity while at work, and the degree to which psoriasis affected activities outside of work. Four scores are derived: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and impairment in activities performed outside of work. Each WPAI score will be expressed as impairment percentages (0-100) with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Percentage of Participants Achieving an sPGA of Clear (0) or Almost Clear (1) with a >=2-Point Decrease from Baseline at Weeks 24, 40, and 52 Comparing TAK-279 Against Apremilast | Baseline, Weeks 24, 40 and 52
  The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scaling, and induration. The average of the 3 scales, rounded to the nearest whole number, is the final sPGA score. The sPGA score ranges from 0 to 4 (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). Higher scores indicate more severe disease activity. 'Clear' and 'Almost clear' will include all participants who score a 0 or 1.
Percentage of Participants Achieving PASI-75 at Weeks 24, 40, and 52 Comparing TAK-279 Against Apremilast | Weeks 24, 40 and 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 75% improvement in PASI score relative to baseline PASI score will be reported.
Percentage of Participants Achieving PASI-90 at Weeks 24, 40, and 52 Comparing TAK-279 Against Apremilast | Weeks 24, 40 and 52
  PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. Percentage of participants showing at least 90% improvement in PASI score relative to baseline PASI score will be reported.
Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESI) | Up to Week 56
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product. An AESI (serious or nonserious) is an adverse event of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator may be appropriate.
Number of Participants with Clinically Significant Vital Signs | Up to Week 56
Number of Participants with Clinically Significant Laboratory Values | Up to Week 56
Number of Participants with Clinically Significant Electrocardiogram (ECG) Findings | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (132):
- United States (27):
  - Saguaro Dermatology Associates, LLC - Probity - PPDS, Phoenix, Arizona
  - First OC Dermatology - Fountain Valley, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - UCLA University of California Los Angeles, Los Angeles, California
  - UC Davis Dermatology Clinic, Sacramento, California
  - Driven Research LLC, Coral Gables, Florida
  - FXM Clinical Research Ft. Lauderdale, LLC, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - FXM Clinical Research Miami, LLC, Miami, Florida
  - Renstar Medical Research -21 NE 1st Ave, Ocala, Florida
  - Marietta Dermatology & The Skin Cancer Center - Marietta, Marietta, Georgia
  - Leavitt Clinical Research - 1542 Elk Creek Dr, Idaho Falls, Idaho
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dawes Fretzin Clinical Research Group-7910 N Shadeland Ave, Indianapolis, Indiana
  - Kindred Hair & Skin Center - CAR, Columbia, Maryland
  - Revival Research Corporation - Michigan - ClinEdge - PPDS, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Henderson Clinical Trials, Henderson, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - ALLCUTIS Research, LLC., Portsmouth, New Hampshire
  - Northwell Health Physician Partners Dermatology at Lake Success - BRANY - PPDS, New York, New York
  - Accellacare of Cary, Cary, North Carolina
  - Bexley Dermatology Research - Probity - PPDS, Bexley, Ohio
  - Clinical Research Center of the Carolinas, LLC, Charleston, South Carolina
  - International Clinical Research-Tennessee LLC, Murfreesboro, Tennessee
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Progressive Clinical Research PA - San Antonio, San Antonio, Texas
- Australia (7):
  - St George Dermatology and Skin Cancer Center - Probity - PPDS, Kogarah, New South Wales
  - The Skin Center - Probity - PPDS, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Brisbane, Queensland
  - Skin Health Institute Inc - Probity - PPDS, Carlton, Victoria
  - Sinclair Dermatology-East Melbourne, East Melbourne, Victoria
  - Alfred Health, Parkville, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (10):
  - Beacon Dermatology - Probity - PPDS, Calgary, Alberta
  - Enverus Medical Research - Probity - PPDS, Surrey, British Columbia
  - CCA Medical Research - Probity - PPDS, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre - Probity - PPDS, Barrie, Ontario
  - Kingsway Clinical Research - Probity - PPDS, Etobicoke, Ontario
  - Guelph Dermatology Research - Probity - PPDS, Guelph, Ontario
  - Mediprobe Research Inc, London, Ontario
  - North Bay Dermatology Center - Probity - PPDS, North Bay, Ontario
  - North York Research Inc. - Probity - PPDS, North York, Ontario
  - Research Toronto - Probity - PPDS, Toronto, Ontario
- China (20):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University - PPDS, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The 1st Affiliated Hospital of Wenzhou Medical University - Nanbaixiang Campus, Wenzhou, Zhejiang
- Germany (4):
  - Hautarztpraxis Mahlow, Blankenfelde-Mahlow, Brandenburg
  - Klinikum Oldenburg AöR, Oldenburg, Lower Saxony
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
- Italy (8):
  - ASL 1 L'Aquila - Presidio Ospedaliero San Salvatore, L’Aquila, Abruzzo
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli - Via Pansini 5, Napoli, Campania
  - IRCCS Az. Osp. Universitaria San Martino- IST, Genoa, Liguria
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico -Via Pace 9, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas, Rozzano, Lombardy
  - IRCCS Policlinico San Donato, San Donato Milanese, Lombardy
  - Presidio Ospedaliero Gaspare Rodolico, Catania, Sicily
  - Azienda Usl Toscana Centro - Firenze, Florence, Tuscany
- Japan (14):
  - Nagoya City University Hospital, Nagoya, Aiti
  - Takagi Dermatological Clinic, Obihiro-Shi, Hokkaidô
  - JR Sapporo Hospital, Sapporo, Hokkaidô
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaidô
  - Fukuoka University Hospital, Fukuoka, Hukuoka
  - Saruwatari Dermatology Clinic, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara-Shi, Kanagawa
  - Jichi Medical University Hospital, Shimotsuke-Shi, Tochigi
  - Teikyo University Hospital, Itabashi-Ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-Ku, Tokyo
  - Tokyo Teishin Hospital, Sumida-Ku, Tokyo
  - Ohyama Dermatology Clinic, Kumamoto
  - Dermatology and Ophthalmology Kume Clinic, Sakaishi, Ôsaka
- Poland (19):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions - Lublin, Lublin, Lublin Voivodeship
  - Dermoklinika-Centrum Medyczne s.c, Lódz, Lódzkie
  - Rheumatology Clinic NZOZ Lecznica MAK-MED, Nadarzyn, Masovian Voivodeship
  - Clinical Best Solutions - Warszawa, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Warszawa - MICS - PPDS, Warsaw, Masovian Voivodeship
  - High-Med Przychodnia Specjalistyczna, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - Klinika Ambroziak - Kosiarzy 9A, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Spólka Komandytowa, Bialystok, Podlaskie Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o. - al. Jana Pawla II 50, Gdansk, Pomeranian Voivodeship
  - Derm-art, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM - Slowackiego, Szczecin, West Pomeranian Voivodeship
  - Centrum Medyczne Bydgoszcz- PRATIA - PPDS, Bydgoszcz
  - Centrum Medyczne PROMED, Krakow
  - Uniwersytecki Szpital Kliniczny im. WAM - Centralny Szpital Weteranow-Lodz-ul. Plac J. Hallera 1, Lodz
- South Korea (15):
  - Pusan National University Hospital, Seogu, Busan Gwangyeogsi
  - Chungnam National University Hospital, Daejeon, Daejeon Gwang'yeogsi
  - Georgia Skin and Cancer Clinic, Savannah, Georgia
  - Chosun University Hospital, Gwangju, Gwangju Gwang'yeogsi
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggido
  - CHA Bundang Medical Center, CHA University - PPDS, Bundang-Gu Seongnam-Si, Gyeonggido
  - Seoul National University Bundang Hospital, Bundang-Gu, Gyeonggido
  - Konkuk University Medical Center, Gwangjin-Gu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Jongno-Gu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seocho-Gu, Seoul Teugbyeolsi
  - Soon Chun Hyang University Hospital Seoul, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Seoul Hospital, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Taiwan (8):
  - National Taiwan University Hospital - Hsin-Chu Branch, Hsinchu
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital-Taipei branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
  - National Taiwan University Hospital, Zhong Zheng Qu

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/c67dd5b3d0534f80